CLINICAL TRIAL: NCT04787601
Title: The Effect Of Cognıtıve-Based Neuromuscular Exercıses On Cognıtıve Functıons And Sportıve Performance In Football Players
Brief Title: The Effect Of Cognitive Training On Sportıve Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nevsehir Haci Bektas Veli University (Other)
Responsible Party: Principal Investigator, Muhammet Ozalp, Lecturer, Nevsehir Haci Bektas Veli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: muhammetlifekinetik
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Healthy
Keywords: cognıtıve-based neuromuscular exercıses; cognıtıve functıons; sportıve performance
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Individuals who meet the inclusion criteria, who volunteered to participate in the study and signed the informed consent form will be divided into two groups, the control group and the study group, by simple random randomization. Experimental group cognitive based neuromuscular exercises + classical training; the control group will only do the classic training. A total of 8-week exercise program will be applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive training (Experimental): Cognitive-based neuromuscular exercises will be applied to the experimental group for a total of 8 weeks.
  Interventions: Other: Exercise; Other: Classic Training
- Control (Other): The control group will only do the classic training.
  Interventions: Other: Classic Training

INTERVENTIONS:
Other: Exercise — Cognıtıve-based neuromuscular exercıses will be applied.
  Arms: Cognitive training
Other: Classic Training — Classic match preparation training

SUMMARY:
The aim of this study is to examine the changes in cognitive performance, coordination, anticipation time, proprioception and pass quality of cognitive-based neuromuscular exercises.

DETAILED DESCRIPTION:
The investigators think that with cognitive-based neuromuscular exercises to be applied to football players, concentration, reflexes, balance, coordination, anticipation time, proprioception and pass quality can be improved. Within the scope of the investigators' study,the investigators think that the positive effects of cognitive-based neuromuscular exercises on executive functions can positively affect athlete performance by contributing to rapid thinking, planning and implementation. In this way, footballers will be able to reach high performances on the field and will become more qualified athletes. In addition, it is predicted that the incidence of injuries in athletes will be minimized by improving the parameters such as anticipation time, balance, coordination, reaction time, and proprioception. If the effectiveness of the exercises is proven, it is aimed to contribute to the literature with objective and evidence-based results in order to include cognitive-based exercises in training programs, which are often overlooked in football training programs.

ELIGIBILITY:
Inclusion Criteria:

* being healthy
* 16-19 years old football players
* footballers who train at least 3 days a week
* agree to participate in the study

Exclusion Criteria:

* who have had an injury in the last 6 months that could affect balance and performance
* orthopedic, neurological or congenital problems

Ages: 16 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Cognitive performance | Change from baseline score at the end of 8 week
  Lumosity is a cognitive training platform developed by containing the results of more than 600 million cognitive training tests from more than 35 million people, which contains the largest data set of human cognitive performance available, either web-based or accessible from a mobile phone application. One test selected for each parameter will be applied and evaluated from the tests that include 6 parameters, namely speed, memory, attention, cognitive flexibility, problem solving and mathematics, in cognitive functions through this program on the computer. Each test will be applied to the participants for the first 2 times to practice, and for the next 3 times to be used as a test score. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Reaction test | change from baseline time at the end of 8 week
  Participants' visual reaction time will be measured in the study. The same working environment will be provided for all participants. During the test, Participants' eyes are focused on the screen and head is 40 cm from the screen. will be kept behind. In the choice reaction time test, there is more than one stimulus and each stimulus requires a different response. Four squares will appear on the computer screen and a different letter will be determined on the keyboard for each square. Whichever of the four squares is lit, the corresponding letter of that square will be asked to be pressed from the keyboard. Participants' reaction times to the stimulus will be recorded by the computer and their Choice Reaction Time averages will be determined.
Coordination test | change from baseline score at the end of 8 week
  The test allows evaluating the coordination of different parts of the body. The researcher throws the ball at a distance of 5 m to the player who is trying to play the ball in turn; The player is asked to play with the chest-foot-head, head-left foot-right foot, foot-chest-head in turn. The researcher calculates the sum of three trials. Unit of measure is 1 point per successful trial
Anticipation time | change from baseline time at the end of 8 week
  The time of anticipation will be calculated by means of computer software by measuring the time during which 10 bubbles seen on the computer monitor descend from top to bottom. The bubbles will first go down in red color, and when it comes to the last balloon, the color will turn green. After 5 retries, 20 repetitions will be made. As soon as the target bubble turns green, it will be asked to press the space key on the computer's keyboard, and the mean duration of the anticipation time error value will be calculated.
Evaluation of Proprioceptive Force Sense | change from baseline score at the end of 8 week
  A pressurized biofeedback device will be used to evaluate the proprioceptive force sensation in both knees. At the beginning of the test, the air-filled pressure bag of the device will be placed under the knee joint and the air pressure will be set to 20 mmHg. Individuals will be asked to perform the maximum voluntary isometric contraction of the M. Quadriceps femoris and 50% of this maximum value will be used in the assessment of proprioceptive force sense. Then, individuals will be asked to contact the M. Quadriceps femoris isometrically until participants reach the calculated proprioceptive force-sensing pressure value by following the device gauge. Single and dual tasks will be required from these processes. The process will be repeated three times and its average will be considered as the test result. High deviation scores indicate a feeling of weak knee joint proprioceptive force, while low deflection scores indicate a good sense of knee joint proprioceptive force.
Loughborough Soccer Passing Test | change from baseline score at the end of 8 week
  LSPT was developed to assess the multifaceted aspect of soccer skill including passing.
Turkey Football Federation Club Injury Card: | through study completion, an average of 6 months
  It consists of information including date of injury, time to return to active sports, injury site, injury type, injury mechanism, diagnostic methods and other details

CONTACTS AND LOCATIONS:
Overall Officials: Muhammet Ozalp, Msc, Principal Investigator — Nevsehir Haci Bektas Veli University
Locations (1):
- Kozaklİ Sport Center, Nevşehir, Kozakli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No